CLINICAL TRIAL: NCT00079872
Title: A Randomized Phase 2 Trial of ALIMTA Plus a Comparator Versus Leucovorin Modulated Fluorouracil Plus a Comparator in First Line Treatment of Locally Advanced or Metastatic Colorectal Cancer
Brief Title: Pemetrexed Plus a Comparator Versus a Combination of 2 Comparators in First-Line Treatment of Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2929; H3E-MC-JMAZ
Record Dates: First submitted 2004-03-17; First posted 2004-03-19 (Estimated); Last update posted 2007-11-06 (Estimated); Status verified 2007-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed

SUMMARY:
In this study, patients will receive either pemetrexed plus irinotecan or 5-fluorouracil (5-FU), leucovorin, and irinotecan.

The purposes of this study are to determine:

* How pemetrexed plus irinotecan compares with 5-FU, leucovorin, and irinotecan in terms of efficacy.
* The safety of pemetrexed plus irinotecan and any side effects that might be associated with it as compared with 5-FU, leucovorin, and irinotecan.
* Whether pemetrexed can help patients with colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

The patient must have:

* Histologic or cytologic diagnosis of adenocarcinoma of the colon or rectum.
* Performance status of 0 to 2 on the ECOG Performance Status Scale.
* Standard postoperative adjuvant radiation therapy for rectal cancer is allowed.
* Locally advanced or metastatic disease.
* Must be 18 years of age.

Exclusion Criteria:

The patient must not have:

* Received prior chemotherapy for advanced disease. Prior adjuvant therapy, including 5-FU, is allowed if it has been more than 12 months since the last treatment.
* Received prior treatment with irinotecan in the adjuvant setting.
* Are unable to take vitamin B12 or folic acid.
* Are unable to interrupt aspirin, other nonsteroidal anti-inflammatory drugs, or COX-2 inhibitors for a 5-day period.
* Have a second primary malignancy except carcinoma in situ of the cervix or nonmelanomatous skin cancer, unless that prior malignancy was diagnosed and definitively treated at least 5 years previously with no subsequent evidence of recurrence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2004-02; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
The primary objective is to compare the antitumor activity of pemetrexed plus a comparator with that of leucovorin modulated 5 FU plus a comparator as measured by tumor response rate for patients with locally advanced or metastatic colorectal cancer

SECONDARY OUTCOMES:
The secondary objectives of the study are as follows:
to assess the following time to event efficacy endpoints for patients in both treatment arms:
overall survival
progression free survival
duration of response
to characterize the quantitative and qualitative toxicities of both treatment arms in this patient population

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- Australia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, NSW, QLD, South Australia, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Woodville
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Frankfurt am Main, Germany
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Krete, Greece
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Amsterdam, Netherlands
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Seville, Spain

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com